CLINICAL TRIAL: NCT01920815
Title: Bicuspid Valve Aortopathy: Feasibility of a Comparative Effectiveness Study
Brief Title: Bicuspid Valve Aortopathy Feasibility Study
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Emory University (Other); University of Colorado, Denver (Other); Baylor College of Medicine (Other); University of California, Los Angeles (Other); Penn State University (Other)
Responsible Party: Principal Investigator, Craig Broberg, Associate Professor, Oregon Health and Science University
Other Study IDs: 1R34HL115032-01A1--BAV; OHSU IRB 8330; 1R34HL115032-01A1 (NIH)
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2018-09

CONDITIONS: Bicuspid Aortic Valve
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Beta blocker therapy: Cohort will consist of those actively taking any beta blocker medication. Observation only.
  Interventions: Other: No interventions
- ARB therapy: Cohort will consist of those actively taking any angiotensin receptor blocker medication. Observation only.
  Interventions: Other: No interventions
- No therapy: Cohort will consist of those not taking either beta blocker nor angiotensin receptor blocker. Observation only.
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions
  Other Names: Observation only

SUMMARY:
In order to determine the effectiveness of medical therapy options to prevent enlargement of the aorta in patients with a bicuspid aortic valve, a randomized study will be planned. This feasibility study will gather accurate data on number needed to screen, changes in medication use over time, and variance of the intended study endpoint.

DETAILED DESCRIPTION:
The study will consider all patients with a bicuspid aortic valve and 1) determine the number of patients needed to be screened for a clinical trial, based on patient eligibility percentages applying specific inclusion and exclusion criteria, 2) for those meeting these criteria, follow changes in and compliance with medical therapy over two years, and 3) in a limited subset of eligible patients, perform MRI at baseline and after 2 years to measure the change in aortic area over time.

ELIGIBILITY:
Inclusion Criteria:

* Bicuspid aortic valve
* Aortic measurement of 35 - 49 mm on prior imaging study

Exclusion Criteria:

* Prior aortic valve or thoracic aortic surgery
* Prior aortic dissection
* Other condition associated with enlarged aorta including Coarctation, Marfans, Turner syndrome, Loeys-Dietz, etc.
* Severe aortic stenosis or regurgitation
* Contraindication to MRI such as claustrophobia or implanted pacer/defibrillator
* Anticipated pregnancy, surgery, or move outside the area within 2 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a bicuspid aortic valve.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-10-04 (Actual)

PRIMARY OUTCOMES:
Change in aortic area measured by MRI | 24 months
  Patients will have a baseline and follow up MRI per a specific protocol to measure area of the ascending thoracic aorta. All measurements will be performed by a core imaging lab

SECONDARY OUTCOMES:
Clinical events involving the aorta, including change in medical therapy | 24 months
  We will observe for any major clinical events over time such as need for surgery, as well as changes in medical therapy over time.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - Oregon Health and Science University, Portland, Oregon
  - Penn State, Hershey, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: No